CLINICAL TRIAL: NCT06452459
Title: Evaluation of Glymphatic Function With MRI
Brief Title: Glymphatic MRI Study
Status: Not yet recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Juan Piantino, Associate Professor, Oregon Health and Science University
Other Study IDs: IT Gadolinium Study
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Other: No interventinon — No intervention is anticipated. This is an observational study.

SUMMARY:
This study aims at identifying neuroimaging markers of glymphatic function in humans.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo MRI without anesthesia
* Calculated GFR greater or equal to 60 mL/min/1.73 m2

Exclusion Criteria:

* Inability to obtain consent
* Subject is incarcerated, pregnant, or lactating or suspects they may be pregnant
* Known allergic or hypersensitivity reactions to gadolinium
* Three or more drug allergies from separate drug classes
* Recent or expected beed for imaging with iodinated contrast
* Contraindications to MRI: claustrophobia, weight greater than maximum MRI scanner capacity, presence of metallic foreign body, or implanted devices not documented as MRI safe
* History of neurosurgical procedure or cervical surgery
* Current use of anticoagulation medications
* Contraindication to lumbar puncture (creatinine or INR elevated above laboratory standard cutoffs)

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Contrast enhancement | 2 weeks
  Measurement of contrast intensity in brain parenchyma

IPD SHARING:
Plan to Share IPD: No